CLINICAL TRIAL: NCT04980755
Title: Body Reprogramming as an Adjunct to Biologic Administration in Patients With Severe Asthma: a Feasibility Study
Brief Title: Adapting Body Reprogramming for Severe Asthma: a Feasibility Study
Acronym: BoBSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Plymouth (Other); Plymouth Marjon University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2109166
Record Dates: First submitted 2021-06-16; First posted 2021-07-28 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-01

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase one (Experimental): Participants will be asked to attend four weekly sessions of Body Reprogramming via group video call.
  Each session will include up to 8 patients and will consist of a 25-30 minute live presentation
  Interventions: Other: Body Reprogramming
- Phase two (Experimental): We anticipate that participant sin phase two will complete the same intervention, but it may be somewhat modified following participant feedback in phase one.
  Interventions: Other: Body Reprogramming

INTERVENTIONS:
Other: Body Reprogramming — An educational intervention originally designed for patients with fibromyalgia.

SUMMARY:
There are many symptoms associated with severe asthma, not all of them related to the lung. These are referred to as extra-pulmonary symptoms and their relationship with quality of life is complex.

Body reprogramming (BR) is a non-drug intervention originally developed for fibromyalgia patients with the aim of improving health and wellbeing in a personalised way, with evidence-based lifestyle changes. The frequency and severity of multiple symptoms in severe asthma is similar to fibromyalgia and the investigators propose that BR may be a suitable non-drug intervention for severe asthma patients who are about to step up drug treatment.

Our study aims are therefore to assess how BR may be suitable for people with severe asthma, and to adapt and optimise the programme for these people. In two phases, severe asthma patients will be recruited via a regional severe asthma clinic at the Royal Devon & Exeter National Health Service (NHS) Trust and invited to take part in a short course of BR. In phase one, patients will be asked to attend four weekly researcher-led sessions of BR via video call and be given practice tasks to report on at the subsequent session. Questionnaires will be completed for the first and last session. At the end of BR, patients will also be invited to take part in a focus group. The data collected will inform development of the programme for phase two, which will involve recruitment of severe asthma patient who are about to start biologic drug treatment for their severe asthma

DETAILED DESCRIPTION:
There are many symptoms associated with severe asthma, not all of them asthma specific (e.g. mental fog, fatigue, unexplained pain), and the relationship between these symptoms and quality of life is complex.

Body reprogramming (BR) is another non-drug intervention originally developed for fibromyalgia patients. BR aims to to improve health and wellbeing in a personalised way, with evidence-based lifestyle changes. The frequency and severity of the non-asthma specific symptoms in severe asthma are similar to those experienced by patients with fibromyalgia. Therefore, the investigators propose that BR may be a suitable non-drug intervention for severe asthma patients who report many non-asthma specific symptoms. This intervention includes optimising knowledge of disease management, physical activity, relaxation and other psychological and biological lifestyle changes which aim to improve wellbeing and mood, and this could lead to better self-management of complex symptoms in asthma patients.

Phase 1 Eligible patients attending a severe asthma service at an Royal Devon and Exeter (RD&E) Hospital will be identified by a health professional familiar to them and invited to take part in the study by post, including a Participant Invitation, Information Leaflet and consent form. The Invitation Letter and Patient Information Leaflet will include instructions to read the material carefully and to bring the consent form with them to their next scheduled clinic appointment.

Participants will be asked to attend four weekly sessions of Body Reprogramming via group video call using Zoom. Each session will include up to 8 patients and will consist of a 25-30 minute live presentation delivered by a researcher from the University of Plymouth. At the end of the presentation, there will be an opportunity to ask questions or raise points of interest. Each session will include a 'practice and report back next week' instruction, and participants will be encouraged to provide written after completing all sessions. feedback before Session topics will include: conceptualising severe asthma, stress and happiness, movement and exercise, and eating and asthma triggers.

Demographics (e.g. age) and clinical data (e.g. current drug treatment) will be collected from participants' hospital notes at the start of the programme. Participants will be asked to complete a series of questionnaires for the first and last weeks of Body Reprogramming. These will be posted to participants and returned to the research team using an enclosed Freepost envelope. Questionnaires will include: the Severe Asthma Questionnaire (SAQ), the General Symptom Questionnaire (GSQ), the Positive And Negative Affect Schedule (PANAS), the Asthma Control Questionnaire. At the end of the course participants will be asked to complete the much shorter General Symptom Questionnaire-Asthma (GSQ-A) instead of the full GSQ. In addition to these questionnaires participants will also be asked to complete and return the Global Rating of Change Questionnaire (GRCQ) and the Friends and Family Test after completing the intervention. These should take no longer than 20 minutes to complete.

Following the course, participants will be invited to attend a focus group with up to 5 other participants via video call or a one to one interview also via video. This time will be used to discuss participants experience of Body Reprogramming, including any problems they may have faced. This will last for up to 2 hours and will be recorded using a voice recorder for transcription and analysis by the research team.

Analysis will include generation of summary statistics and mean differences for numerical data, including the number of people who were invited and attended each BR course.

Thematic analysis of transcribed focus group data will be used to inform any changes which need to made to improve the programme before Phase 2.

Phase 2 Before commencing a biologic treatment for severe asthma in normal clinic care, patients are reviewed by a multidisciplinary team responsible for their care, and the participating hospital's Principal Investigator will identify eligible participants. Participant recruitment will then proceed as outlined in Phase 1.

A modified GRCQ will completed by participants at the end of the intervention in phase 2. The changes to the wording of GRCQ are to take into account that participants have started a new treatment (the biologic drug) and completed BR. Except for this change, the same questionnaire data will be collected at the same time-points in this phase.

ELIGIBILITY:
Inclusion Criteria:

* Phase one:

  * Aged ≥18 years attending the regional specialist severe asthma service in Royal Devon and Exeter hospitals.
  * Diagnosed with severe asthma as per European Respiratory Society/American Thoracic Society (ERS/ATS) definition.

    * Requiring high dose inhaled corticosteroids (NICE definition of high dose ICS).
  * Eight or more non-respiratory symptoms per week (approximately 60% of patients with severe asthma have a moderate or high extra-pulmonary symptom burden) as measured by the General Symptom Questionnaire
* Phase two:

  * Diagnosed with severe asthma as per ERS/ATS definition.

    * Requiring high dose inhaled corticosteroids (NICE definition of high dose ICS).
  * Patients with severe asthma who have been approved for biologic treatment according to national guidance and have been assessed by a multi-disciplinary team will be offered the intervention pending starting their biologic treatment.
  * Patients with eight or more non-respiratory symptoms per week as measured by the GSQ.

Exclusion Criteria:

* Phase one and Phase two

  * Unable or unwilling to partake.
  * In the opinion of the patient's treating physician, the patient has another condition which is significantly impairs their ability to take part in the BR.
  * No access to the internet or appropriate IT equipment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Masoli, MD, Principal Investigator — Royal Devon and Exeter Hopsitals NHS Trust
Locations (1):
- Royal Devon and Exeter Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Enrolled in Body Reprogramming: Patients enrolled in one of the Body Reprogramming courses
Period: Body Reprogramming Courses
Arm/Group | Patients Enrolled in Body Reprogramming
Started | 28
Completed | 13
Not Completed | 15
Not completed — Too unwell to attend | 6
Not completed — Work commitment | 2
Not completed — Unsure when the course started | 1
Not completed — Could not be contacted to provide a reason | 6
Period: Post-course Interviews
Arm/Group | Patients Enrolled in Body Reprogramming
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: Years] | 50 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 26
  Mixed race | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Taking Part Who Completed All 4 Weeks of the Course
Description: Consistent course attendance with the course will be used to infer participants level of engagement with the course content. Reasons for consistent attendance, or poor attendance, will be explored further with participants during the semi-structured interviews.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 28
Participants | 13

2. Primary Outcome: Number and Percentage of Participants Who Complete the Study Questionnaires
Description: By capturing this information, we will determine if one of our study questionnaires is routinely unfinished by the study participants. Reasons for this can be explored during the focus groups or one to one interviews.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 28
Participants | 16

3. Primary Outcome: Number and Percentage of Participants Who Complete the Study Questionnaires
Description: See outcome 2
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 13
Participants | 8

4. Secondary Outcome: Number of Participants Who Attended Two or More Sessions and Were Invited to a Follow-up Interview
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 28
Participants | 19

5. Secondary Outcome: Of Those Invited, the Number Who Accepted an Invitation to Take Part in a Follow-up Interview
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Enrolled in Body Reprogramming
Number analyzed (Participants) | 19
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed
Description: Adverse events were not monitored/assessed. This study concerned a low burden, educational intervention. No changes were made to the participants' medications, and no adverse events were anticipated or monitored in the context of this study
Arm/Group | Patients Enrolled in Body Reprogramming
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT04980755/Prot_SAP_000.pdf